CLINICAL TRIAL: NCT01498068
Title: Open-Label, Bridging Study to Determine Efficacy and Safety of Telaprevir, Pegylated-Interferon-alfa-2a and Ribavirin in Treatment- Naïve and Treatment-Experienced Russian Subjects With Genotype 1 Chronic Hepatitis C
Brief Title: Open-Label, Bridging Study of Telaprevir in Treatment-Naïve and Treatment-Experienced Russian Patients With Genotype 1 Chronic Hepatitis C
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR100676; VX-950HPC3007 (Other: Janssen-Cilag International NV, Belgium)
Record Dates: First submitted 2011-12-06; First posted 2011-12-23 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Genotype 1 Chronic Hepatitis C
Keywords: Genotype 1 chronic Hepatitis C; VX-950HPC3007; VX-950; Hepatitis C; Telaprevir; HCV
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment-naïve (Experimental): Treatment naïve participants will receive telaprevir 750 mg 8 hourly for 12 weeks in combination with Peg-IFN alfa-2a 180 microgram weekly and RBV 1000 - 1200 mg daily (dependent on weight) for 24 or 48 weeks. Total treatment duration will be based on participant's prior treatment status, liver disease status, and individual ontreatment virologic response in this study.
  Interventions: Drug: Telaprevir; Drug: Pegylated-interferon-alfa-2a; Drug: Ribavirin
- Treatment-experienced (Experimental): Treatment-experienced participants received telaprevir 750 mg 8 hourly for 12 weeks in combination with Peg-IFN alfa-2a 180 microgram weekly and RBV 1000 - 1200 mg daily (dependent on weight) for 24 or 48 weeks. Total treatment duration will be based on participant's prior treatment status, liver disease status, and individual on-treatment virologic response in this study.
  Interventions: Drug: Telaprevir; Drug: Pegylated-interferon-alfa-2a; Drug: Ribavirin

INTERVENTIONS:
Drug: Telaprevir — Telaprevir Type = exact number, unit = mg, number = 750, form = tablet, route = oral. Telaprevir 750 mg (2 oral tablets) is taken every 8 hours for 12 weeks
Drug: Pegylated-interferon-alfa-2a — Pegylated-interferon-alfa-2a type = exact number, unit = microgram, number = 180, form = injection, route = subcutaneous. 180 microgram (µg) per week, subcutaneous injection, for 24 or 48 weeks
Drug: Ribavirin — Ribavirin Type = exact, number = 1000 or 1200, unit = mg, form = tablet, route = oral. 1000mg (if participant's weight is < 75kg) or 1200mg (if participant's weight is >= 75kg) per day for 24 or 48 weeks.

SUMMARY:
The purpose of this study is to determine the effectiveness, safety and tolerability of telaprevir administered as 750 mg every 8 hours (q8h) in combination with pegylated interferon (Peg-IFN)-alfa-2a and ribavirin (RBV) in treatment-naïve and treatment-experienced Russian participants with genotype 1 chronic hepatitis C.

DETAILED DESCRIPTION:
This is an open-label (all persons know the study drug assignment), multicenter study in treatment-naïve (participant did not receive any previous treatment for the treatment of hepatitis C) and treatment-experienced (participant did receive previous treatment for hepatitis C) Russian participants with genotype 1 chronic hepatitis C. After a screening period of approximately 4 weeks, participants will be treated for 12 weeks with telaprevir 750 mg every 8 hours in combination with Peg-IFN-alfa-2a and RBV followed by 12 or 36 weeks of treatment with Peg-IFN-alfa-2a and RBV alone depending on their liver disease status, response to previous treatment and individual virologic response during treatment in this study. After the treatment period, there is a follow-up phase of at least 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participant has genotype 1 chronic hepatitis C with HCV RNA level >1000 IU/mL
* Participant is either treatment-naïve and did not receive any previous treatment with any approved or investigational drug or drug regimen for the treatment of hepatitis C, or participant is treatment-experienced who did not achieve sustained virologic response (SVR) 24 weeks after at least 1 prior course of Peg-IFN/RBV therapy (null-responder, partial-responder or viral relapse)
* Participant must have documentation of liver biopsy or fibroscan within 2 years before the screening visit or agree to have a biopsy or fibroscan within the screening period unless histological cirrhosis was demonstrated by a biopsy or fibroscan > 2 years ago prior to screening
* A female participant of childbearing potential and a nonvasectomized male participant who has a female partner of childbearing potential must agree to the use of 2 effective methods of birth control from screening until 6 months (female participant ) or 7 months (male participant) after the last dose of RBV

Exclusion Criteria:

* Prior non-responder that is classified as a viral breakthrough participant
* Participant is infected or co-infected with HCV of another genotype than genotype 1
* Participant has history of decompensated liver disease or shows evidence of significant liver disease in addition to hepatitis C
* Participant has human immunodeficiency virus (HIV) or hepatitis B virus (HBV) co-infection
* Participant has active malignant disease or history of malignant disease within the past 5 years (with the exception of treated basal cell carcinoma or hepatocellular carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV, Belgium Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (5):
- Russia (5):
  - Moscow
  - Saint Petersburg
  - Samara
  - Smolensk
  - Stavropol

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 sites in Russia.
Pre-assignment Details: Of the 39 participants screened, 36 participants (16 treatment-naïve/ 20 treatment-experienced) were enrolled and treated.
Groups:
- Treatment-naïve: Treatment naïve participants received telaprevir 750 mg every 8 hours for 12 weeks in combination with Peg-IFN alfa-2a 180 microgram once a week and RBV 1000 - 1200 mg daily (dependent on weight) for 24 or 48 weeks. Total treatment duration is based on participant's prior treatment status, liver disease status, and individual on-treatment virologic response in this study.
- Treatment-experienced: Treatment-experienced participants received telaprevir 750 mg every 8 hours for 12 weeks in combination with Peg-IFN alfa-2a 180 microgram once a week and RBV 1000 - 1200 mg daily (dependent on weight) for 24 or 48 weeks. Total treatment duration is based on participant's prior treatment status, liver disease status, and individual on-treatment virologic response in this study.
Period: Overall Study
Arm/Group | Treatment-naïve | Treatment-experienced
Started | 16 | 20
Completed | 15 | 19
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-naïve | Treatment-experienced | Total
Number analyzed (Participants) | 16 | 20 | 36
Age, Customized [Number; unit: Participants]
  <= 45 years | 13 | 12 | 25
  Between 45 and 65 years | 2 | 8 | 10
  > 65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Extended Rapid Virologic Response (eRVR)
Description: A eRVR is defined as having hepatitis C virus (HCV) ribonucleic acid (RNA) less than 25 IU/mL, (target not detected) at Weeks 4 and 12 of treatment.
Time Frame: Week 4 and Week 12
Population: Full analysis (FA) population: All participants who received at least one dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Treatment-naïve | Treatment-experienced
Number analyzed (Participants) | 16 | 20
Participants | 13 | 18

2. Secondary Outcome: Median Change in log10 Hepatitis C Virus (HCV) Ribonucleic Acid (RNA)
Description: Changes from baseline in log10 HCV RNA levels were calculated.
Time Frame: Baseline (Week 0), Week 4, Week 8, Week 12, Week 24, Week 32, Week 40, and Week 48
Population: Full analysis (FA) population: All participants who received at least one dose of the study medication. "n" signifies number of participants who were evaluable at each specified timepoint for each arm, respectively.
Measure: Median (Full Range); unit: Log 10 IU/mL
Arm/Group | Treatment-naïve | Treatment-experienced
Number analyzed (Participants) | 16 | 20
Log 10 IU/mL
  Baseline (n=16, 20) | 6.20 [4.6 to 6.9] | 6.10 [5.7 to 7.0]
  Week 4 (n=16, 20) | -5.47 [-6.2 to -3.9] | -5.33 [-6.3 to -3.5]
  Week 8 (n=16,19) | -5.50 [-6.2 to -3.9] | -5.39 [-6.3 to -5.00]
  Week 12 (n=15,19) | -5.46 [-6.2 to -3.9] | -5.39 [-6.3 to -5.00]
  Week 24 (n=14, 19) | -5.53 [-6.2 to -3.9] | -5.39 [-6.3 to -0.6]
  Week 32 (n=2, 12) | -5.30 [-5.5 to -5.1] | -5.46 [-6.3 to -5.2]
  Week 40 (n=2, 12) | -5.30 [-5.5 to -5.1] | -5.46 [-6.3 to -5.2]
  Week 48 (n=2, 12) | -3.14 [-5.1 to -1.2] | -5.46 [-6.3 to -5.2]

3. Secondary Outcome: Number of Participants With Rapid Virologic Response (RVR) at Week 4
Description: A RVR is defined as having hepatitis C virus (HCV) ribonucleic acid (RNA) less than 25 IU/mL, (target not detected) at Week 4
Time Frame: Week 4
Population: Full analysis (FA) population: All participants who received at least one dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Treatment-naïve | Treatment-experienced
Number analyzed (Participants) | 16 | 20
Participants | 14 | 18

4. Secondary Outcome: Number of Participants With Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Less Than 25 IU/mL, (Target Not Detected) at Weeks 8, 12, 24, 32, 40 and 48
Description: The table below shows number of participants with HCV RNA Less than 25 IU/mL, (target not detected) at Weeks 8, 12, 24, 32, 40 and 48. Only 3 treatment-naive and 14 Treatment-experienced participants were assigned to receive study treatment after Week 24. Only participants still receiving Treatment were assessed at 32, 40, and 48 weeks.
Time Frame: Weeks 8, 12, 24, 32, 40 and 48
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | Treatment-naïve | Treatment-experienced
Number analyzed (Participants) | 16 | 20
Participants
  Week 8 (n=16, 20) | 16 | 19
  Week 12 (n=16, 20) | 15 | 19
  Week 24 (n=16, 20) | 15 | 18
  Week 32 (n=3, 14) | 2 | 12
  Week 40 (n=3, 14) | 2 | 12
  Week 48 (n=3, 14) | 1 | 12

5. Secondary Outcome: Number of Participants With Virologic Failure
Description: Virologic failure is defined as hepatitis C virus (HCV) ribonucleic acid (RNA) levels more than 1,000 IU/mL at Weeks 4, 8, 12, 24, 32, or 40.
Time Frame: Week 4, Week 8, Week 12, Week 24, Week 32, or Week 40
Population: Full analysis (FA) population: All participants who received at least one dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Treatment-naïve | Treatment-experienced
Number analyzed (Participants) | 16 | 20
Participants | 1 | 2

6. Secondary Outcome: Number of Participants in Each Specific Category of Treatment Outcome
Description: Participants were evaluated for following 4 categories of treatment outcome;Sustained Virologic Response 12 Weeks After Last Planned Dose of Study Medication(SVR12):hepatitis C virus (HCV)ribonucleic acid (RNA)<25 IU/mL(target not detected)12 weeks after last planned dose of study medication;Relapse:HCV RNA =>25 IU/mL during follow-up period after previous HCV RNA<25 IU/mL at planned end of treatment(EOT)[Week 24 or Week 48] and participant did not achieve SVR12planned;On treatment virologic failure:meeting virologic stopping rule and/or having detectable HCV RNA at EOT with viral breakthrough(having a confirmed increase >1 log 10 in HCV RNA level from the lowest level reached or confirmed value of HCV RNA >100 IU/mL in participants whose HCV RNA has previously become <25 IU/mL during treatment).Stopping rule defined as HCV RNA value >1000 IU/mL at Week 4, 8 or 12 or detectable HCV RNA at Week 24, 32 or 40;Other:HCV RNA <25 IU/mL at actual EOT and never HCV RNA =>25 IU/mL thereafter.
Time Frame: From Day 1 (Baseline) up to Follow-up visit (Week 36 or Week 60)
Population: Full analysis (FA) population: All participants who received at least one dose of the study medication.
Measure: Number; unit: Participants
Arm/Group | Treatment-naïve | Treatment-experienced
Number analyzed (Participants) | 16 | 20
Participants
  SVR12 | 14 | 16
  Relapse | 0 | 1
  On treatment virologic failure | 1 | 2
  Other | 1 | 1

ADVERSE EVENTS:
Time Frame: 60 weeks
Arm/Group | Treatment-naïve | Treatment-experienced
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/20
Other Adverse Events (participants affected / at risk) | 16/16 | 19/20
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naïve (N=16) | Treatment-experienced (N=20)
Influenza like illness (General disorders) | 6 | 9
Pyrexia (General disorders) | 6 | 3
Anaemia (Blood and lymphatic system disorders) | 6 | 6
Neutropenia (Blood and lymphatic system disorders) | 2 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Alanine aminotransferase increased (Investigations) | 2 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Anal pruritus (Gastrointestinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Injection site erythema (General disorders) | 1 | 1
Asthenia (General disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days